CLINICAL TRIAL: NCT02378714
Title: Behavioral Activation and Varenicline for Smoking Cessation in Depressed Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brian Hitsman, Associate Professor of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00100303; 1R01CA184211-01A1 (NIH)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-05

CONDITIONS: Nicotine Dependence; Major Depressive Disorder
Keywords: Smoking Cessation; Major Depressive Disorder; Nicotine Dependence; Varenicline; Behavioral Activation Therapy; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Depressive Disorder, Major; Smoking Cessation; Cigarette Smoking | interventions — Varenicline; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard treatment + placebo varenicline (Placebo Comparator): Standard behavioral smoking cessation treatment plus placebo varenicline
  Interventions: Behavioral: Standard treatment
- BASC + placebo varenicline (Experimental): Behavioral activation for smoking cessation plus placebo varenicline
  Interventions: Behavioral: BASC
- Standard treatment + active varenicline (Active Comparator): Standard behavioral smoking cessation treatment plus active varenicline
  Interventions: Drug: Varenicline; Behavioral: Standard treatment
- BASC + active varenicline (Experimental): Behavioral activation for smoking cessation plus active varenicline
  Interventions: Drug: Varenicline; Behavioral: BASC

INTERVENTIONS:
Drug: Varenicline — Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
  Other Names: Chantix
  Arms: BASC + active varenicline; Standard treatment + active varenicline
Behavioral: BASC — The goal of behavioral activation therapy is to increase engagement in rewarding activities, a problem for smokers with depression who find smoking especially rewarding and prefer it over many other traditionally rewarding activities, by reducing patterns of behavioral avoidance, withdrawal, and inactivity. In this study, behavioral activation will be integrated with standard behavioral smoking cessation treatment.
  Treatment will be delivered in eight 45-minute sessions over 12 weeks occurring weekly for the first four sessions and biweekly for the final four sessions.
  Other Names: Behavioral activation for smoking cessation
  Arms: BASC + active varenicline; BASC + placebo varenicline
Behavioral: Standard treatment — Standard behavioral smoking cessation treatment is an effective treatment for nicotine dependence. Treatment focuses on self-monitoring of smoking behavior, identifying smoking triggers and alternative trigger management strategies, relaxation, social support for non-smoking, and relapse prevention. Treatment will be delivered in eight 45-minute sessions over 12 weeks occurring weekly for the first four sessions and biweekly for the final four sessions.
  Other Names: Standard Therapy
  Arms: Standard treatment + active varenicline; Standard treatment + placebo varenicline

SUMMARY:
Persons who struggle with depression smoke at high rates and experience low quit rates in treatment. The best way to improve cessation treatment for this underserved population remains unknown. The proposed trial tests whether the combination of varenicline and behavioral mood management treatment enhances long-term abstinence for depressed smokers and, if so, whether this treatment achieves its effects through addressing the unique psychological factors that appear to maintain tobacco dependence for these smokers.

DETAILED DESCRIPTION:
Upwards of 43% of persons with major depressive disorder (MDD) are daily smokers who are more likely to smoke heavily, show greater tobacco dependence, suffer more severe withdrawal, and experience lower quit rates than smokers without MDD. Little is known about treatment strategies that might optimize smoking cessation for smokers with MDD because almost all randomized clinical trials have excluded these smokers. This project answers many prominent but largely unanswered calls over the last decade to address tobacco dependence in persons with mental health disorders, especially major depressive disorder (MDD). Using a double-blind, placebo-controlled, randomized design, the investigators will evaluate the efficacy of behavioral activation for smoking cessation (BASC) plus varenicline for treating tobacco dependence in smokers with current or lifetime MDD. Three hundred and thirty daily (≥1 cigarettes/day) smokers will be randomized to receive 12 weeks of one of four treatments: 1) Standard behavioral cessation treatment (ST) + placebo; 2) Behavioral activation integrated with ST (BASC) + placebo; 3) ST + varenicline; or 4) BASC + varenicline. Both BASC and ST will be administered in eight 45 minute sessions, occurring weekly for the first four weeks and biweekly for the final eight weeks. Randomization will be stratified on clinical site (Northwestern, University of Pennsylvania), gender, and severity of depressive symptoms (minimal/mild vs. moderate/severe). The primary outcomes will be carbon monoxide (CO) verified 7-day point prevalence abstinence at 24-weeks post-quit. Additional aims include assessing adverse event rates between varenicline and placebo arms, and testing for mediation of treatment effects by anhedonia, cognitive function (attention and memory), cigarette reward value, and craving and withdrawal. This randomized controlled trial will be the first adequately powered trial of BASC in this population; the first trial to evaluate varenicline among a community sample of smokers with MDD; and the first trial to assess the main and combined effects of these two treatments.

ELIGIBILITY:
Inclusion criteria:

1. adult (18 years of age or older) daily cigarette smokers (1+ cigarettes per day)
2. meet criteria for current or lifetime MDD without psychotic features
3. have or are willing to acquire a personal email address and access to a camera phone or other method for submission of therapy practice assignments
4. speak, read, and write fluently in English
5. able to provide written informed consent
6. intend to reside in the geographic area for >8 months
7. women of childbearing potential must agree to use a medically acceptable method of birth control or abstain from sexual intercourse during the time they are taking study medication and for at least one month after the medication period ends.
8. The candidate had to answer "yes" to the question: "Are you interested in quitting smoking?"

Exclusion criteria:

1. current enrollment or plan to enroll in another smoking cessation program in the next 8 months
2. regular (daily) use of e-cigarettes, chewing tobacco, snuff, snus, or other tobacco products
3. current use or plan to use nicotine replacement therapy or other smoking cessation medication within the next 8 months
4. medications indicated for bipolar or psychotic disorder if prescribed for bipolar or psychotic disorder
5. pregnant or planning to become pregnant within the next 8 months, or breast feeding
6. history of seizures or current seizure disorder without medication
7. history of severe (stage IV or V) chronic kidney disease including current or prior end stage renal disease on either hemodialysis or peritoneal dialysis or prior renal transplant
8. any prior solid organ transplant or prior hematopoietic stem cell transplant
9. alcohol consumption exceeding 28 drinks per week
10. cirrhosis or end-stage liver disease
11. systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg after two readings or symptomatic uncontrolled stage II hypertension
12. unstable cardiovascular disease within 3 months prior to baseline or other cardiovascular disease requiring hospitalization
13. prior hospitalization for heart failure
14. previous allergic reaction to varenicline
15. high suicide risk based on the Columbia Suicide Severity Rating Scale
16. lifetime bipolar or psychotic disorder as determined by either self-report or clinical interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hitsman, Ph.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Anthenelli RM, Morris C, Ramey TS, Dubrava SJ, Tsilkos K, Russ C, Yunis C. Effects of varenicline on smoking cessation in adults with stably treated current or past major depression: a randomized trial. Ann Intern Med. 2013 Sep 17;159(6):390-400. doi: 10.7326/0003-4819-159-6-201309170-00005. PMID 24042367
- [Background] Blalock JA, Robinson JD, Wetter DW, Schreindorfer LS, Cinciripini PM. Nicotine withdrawal in smokers with current depressive disorders undergoing intensive smoking cessation treatment. Psychol Addict Behav. 2008 Mar;22(1):122-8. doi: 10.1037/0893-164X.22.1.122. PMID 18298238
- [Background] Ebbert JO, Wyatt KD, Hays JT, Klee EW, Hurt RD. Varenicline for smoking cessation: efficacy, safety, and treatment recommendations. Patient Prefer Adherence. 2010 Oct 5;4:355-62. doi: 10.2147/ppa.s10620. PMID 21049087
- [Background] Gierisch JM, Bastian LA, Calhoun PS, McDuffie JR, Williams JW Jr. Smoking cessation interventions for patients with depression: a systematic review and meta-analysis. J Gen Intern Med. 2012 Mar;27(3):351-60. doi: 10.1007/s11606-011-1915-2. Epub 2011 Oct 26. PMID 22038468
- [Background] Hitsman B, Moss TG, Montoya ID, George TP. Treatment of tobacco dependence in mental health and addictive disorders. Can J Psychiatry. 2009 Jun;54(6):368-78. doi: 10.1177/070674370905400604. PMID 19527557
- [Background] Hitsman B, Papandonatos GD, McChargue DE, DeMott A, Herrera MJ, Spring B, Borrelli B, Niaura R. Past major depression and smoking cessation outcome: a systematic review and meta-analysis update. Addiction. 2013 Feb;108(2):294-306. doi: 10.1111/add.12009. PMID 23072580
- [Background] Philip NS, Carpenter LL, Tyrka AR, Whiteley LB, Price LH. Varenicline augmentation in depressed smokers: an 8-week, open-label study. J Clin Psychiatry. 2009 Jul;70(7):1026-31. doi: 10.4088/jcp.08m04441. Epub 2009 Mar 24. PMID 19323966
- [Background] MacPherson L, Tull MT, Matusiewicz AK, Rodman S, Strong DR, Kahler CW, Hopko DR, Zvolensky MJ, Brown RA, Lejuez CW. Randomized controlled trial of behavioral activation smoking cessation treatment for smokers with elevated depressive symptoms. J Consult Clin Psychol. 2010 Feb;78(1):55-61. doi: 10.1037/a0017939. PMID 20099950
- [Derived] Gollan JK, Liverant G, Jao NC, Lord KA, Whitton AE, Hogarth L, Fox E, Bauer AM, Quinn MH, Pizzagalli DA, Leone FT, Papandonatos GD, Schnoll RA, Hitsman B. Depression Severity Moderates Reward Learning Among Smokers With Current or Past Major Depressive Disorder in a Smoking Cessation Randomized Clinical Trial. Nicotine Tob Res. 2024 Apr 22;26(5):639-644. doi: 10.1093/ntr/ntad221. PMID 37943674
- [Derived] Schnoll R, Wileyto EP, Bauer AM, Fox EN, Blumenthal D, Hosie Quinn M, Leone F, Huffman MD, Khan SS, Gollan JK, Papandonatos GD, Hitsman B. Seeing Through the Blind: Belief About Treatment Randomization and Smoking Cessation Outcome Among People With Current or Past Major Depressive Disorder Who Smoke in a Placebo-Controlled Trial of Varenicline. Nicotine Tob Res. 2024 Apr 22;26(5):597-603. doi: 10.1093/ntr/ntad218. PMID 37934573
- [Derived] Carroll AJ, Huffman MD, Wileyto EP, Khan SS, Fox E, Smith JD, Bauer AM, Leone FT, Schnoll RA, Hitsman B. Change in cardiovascular health among adults with current or past major depressive disorder enrolled in intensive smoking cessation treatment. J Affect Disord. 2023 Jul 15;333:527-534. doi: 10.1016/j.jad.2023.04.089. Epub 2023 Apr 28. PMID 37119868
- [Derived] Hitsman B, Papandonatos GD, Gollan JK, Huffman MD, Niaura R, Mohr DC, Veluz-Wilkins AK, Lubitz SF, Hole A, Leone FT, Khan SS, Fox EN, Bauer AM, Wileyto EP, Bastian J, Schnoll RA. Efficacy and safety of combination behavioral activation for smoking cessation and varenicline for treating tobacco dependence among individuals with current or past major depressive disorder: A 2 x 2 factorial, randomized, placebo-controlled trial. Addiction. 2023 Sep;118(9):1710-1725. doi: 10.1111/add.16209. Epub 2023 May 3. PMID 37069490
- See also: FDA Product Information for Varenicline — http://www.accessdata.fda.gov/drugsatfda_docs/label/2009/021928s012s013lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- BASC + Placebo Varenicline: Behavioral activation for smoking cessation plus placebo varenicline
  BASC: The goal of behavioral activation therapy is to increase engagement in rewarding activities, a problem for smokers with depression who find smoking especially rewarding and prefer it over many other traditionally rewarding activities, by reducing patterns of behavioral avoidance, withdrawal, and inactivity. In this study, behavioral activation will be integrated with standard behavioral smoking cessation treatment.
  Treatment will be delivered in eight 45-minute sessions over 12 weeks occurring weekly for the first four sessions and biweekly for the final four sessions.
- BASC + Active Varenicline: Behavioral activation for smoking cessation plus active varenicline
  Varenicline: Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
  BASC: The goal of behavioral activation therapy is to increase engagement in rewarding activities, a problem for smokers with depression who find smoking especially rewarding and prefer it over many other traditionally rewarding activities, by reducing patterns of behavioral avoidance, withdrawal, and inactivity. In this study, behavioral activation will be integrated with standard behavioral smoking cessation treatment.
  Treatment will be delivered in eight 45-minute sessions over 12 weeks occurring weekly for the first four sessions and biweekly for the final four sessions.
Period: Overall Study
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Started | 68 | 68 | 81 | 83
Completed | 39 | 29 | 51 | 51
Not Completed | 29 | 39 | 30 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline | Total
Number analyzed (Participants) | 68 | 68 | 81 | 83 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 63 | 58 | 74 | 75 | 270
  >=65 years | 5 | 10 | 7 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.8) | 50.7 (13.5) | 48.7 (12.7) | 50.3 (13.2) | 50.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 44 | 44 | 165
  Male | 29 | 30 | 37 | 39 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 40 | 37 | 43 | 37 | 157
  White | 25 | 27 | 28 | 36 | 116
  More than one race | 1 | 3 | 4 | 8 | 16
  Unknown or Not Reported | 2 | 0 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 68 | 68 | 81 | 83 | 300

OUTCOME MEASURES:

1. Primary Outcome: Bioverified Point-prevalence Abstinence at 27 Weeks
Description: Participants were classified as abstinent if they reported abstinence, not even a puff of a cigarette, for >7 days prior to week 27 (24 weeks post-target quit date) and had an expired carbon monoxide reading of ≤ 6 parts per million at week 27.
Time Frame: 27 weeks (24-weeks post-target quit date)
Population: All participants enrolled in the trial (intent-to-treat sample)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Number analyzed (Participants) | 68 | 68 | 81 | 83
Participants | 6 | 3 | 13 | 13

2. Primary Outcome: Adverse Event and Serious Adverse Event Rates
Description: Adverse event and serious adverse event rates between varenicline and placebo arms. A previously developed algorithm was used to classify side effect reports as adverse events (AEs) or serious adverse events (SAEs) (Schnoll et al. 2019).
  Reference: Schnoll, R., Leone, F., Weisbrot, J., Veluz-Wilkins, A., Miele, A., Hole, A., Jao, N.C., Wileyto, E.P., Carroll, A.J., Kalhan, R., Patel, J., Langer, C., & Hitsman, B. (2019). A randomized controlled trial of 24-weeks of varenicline for tobacco use among cancer patients: Efficacy, safety, and adherence. Psycho-Oncology, 28, 561-569.
Time Frame: Weeks 1 (1-week before starting medication), 6, and 14 (end of medication)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Week 1: Placebo group during first week of treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 1: Varenicline group during first week of treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 6; Varenicline - Week 6: Placebo group mid-treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 14; Varenicline - Week 14: Placebo group at end of treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
Arm/Group | Placebo - Week 1 | Varenicline - Week 1 | Placebo - Week 6 | Varenicline - Week 6 | Placebo - Week 14 | Varenicline - Week 14
Number analyzed (Participants) | 136 | 164 | 91 | 121 | 74 | 104
Participants
  Any adverse event | 104 | 136 | 68 | 81 | 50 | 60
  Any serious adverse event | 28 | 34 | 26 | 22 | 9 | 8

3. Secondary Outcome: Bioverified Point-prevalence Abstinence at 14 Weeks (End of Treatment)
Description: Participants were classified as abstinent if they reported abstinence, not even a puff of a cigarette, for >7 days prior to week 14 (11-weeks post-target quit date) and had an expired carbon monoxide reading of ≤ 6 parts per million at week 14.
Time Frame: 14 weeks (11-weeks post-target quit date)
Population: All participants enrolled in the trial (intent-to-treat sample)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Number analyzed (Participants) | 68 | 68 | 81 | 83
Participants | 8 | 4 | 26 | 26

4. Secondary Outcome: Prolonged Abstinence
Description: <7 consecutive days of self-reported smoking after a 2-week grace period
Time Frame: 27 weeks (24 weeks post target quit date)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Number analyzed (Participants) | 57 | 45 | 68 | 70
Participants | 13 | 11 | 26 | 26

5. Secondary Outcome: Continuous Abstinence
Description: No smoking between target quit date (week 3) and week 27
Time Frame: 27 weeks (24 weeks post target quit date)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Number analyzed (Participants) | 59 | 52 | 72 | 71
Participants | 3 | 2 | 6 | 2

6. Secondary Outcome: Time to 7-day Relapse
Description: Time to relapse as defined by 7 or more consecutive days of self-reported smoking (no grace period)
Time Frame: 27 weeks (24 weeks post target quit date)
Measure: Median (95% Confidence Interval); unit: median days to relapse
Arm/Group | Standard Treatment + Placebo Varenicline | BASC + Placebo Varenicline | Standard Treatment + Active Varenicline | BASC + Active Varenicline
Number analyzed (Participants) | 57 | 45 | 68 | 70
median days to relapse | 15 [15 to 16] | 15 [15 to 22] | 57 [15 to 144] | 24 [15 to 135]

ADVERSE EVENTS:
Time Frame: Medication side effects were measured using a 28-item side effect checklist rating scale at week 1 (1 week before starting medication), week 3 (target quit day) through 14, and week 27.
Description: Adverse events and serious adverse events are reported only for active and placebo medication arms, which aligns with our primary aim for varenicline safety and the statistical analysis plan.
Groups:
- Placebo - Week 3: Placebo group at week 3.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 3: Varenicline group at week 3.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 4: Placebo group at week 4.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 4: Varenicline group at week 4.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 6: Varenicline group mid-treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 7: Placebo group at week 7.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 7: Varenicline group at week 7.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 8: Placebo group at week 8.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 8: Varenicline group at week 8.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 10: Placebo group at week 10.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 10: Varenicline group at week 10.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 12: Placebo group at week 12.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 12: Varenicline group at week 12.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 14: Varenicline group at end of treatment.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Placebo - Week 27: Placebo group at week 27.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
- Varenicline - Week 27: Varenicline group at week 27.
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Participants will be randomly assigned to 12 weeks of either placebo or varenicline medication (1mg twice daily). Participants and research personnel will be blind to treatment assignment.
Arm/Group | Placebo - Week 1 | Varenicline - Week 1 | Placebo - Week 3 | Varenicline - Week 3 | Placebo - Week 4 | Varenicline - Week 4 | Placebo - Week 6 | Varenicline - Week 6 | Placebo - Week 7 | Varenicline - Week 7 | Placebo - Week 8 | Varenicline - Week 8 | Placebo - Week 10 | Varenicline - Week 10 | Placebo - Week 12 | Varenicline - Week 12 | Placebo - Week 14 | Varenicline - Week 14 | Placebo - Week 27 | Varenicline - Week 27
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/164 | 0/114 | 0/137 | 0/100 | 0/120 | 0/91 | 0/121 | 0/85 | 0/119 | 0/80 | 0/115 | 0/79 | 0/113 | 0/79 | 0/109 | 0/74 | 0/104 | 0/68 | 0/102
Serious Adverse Events (participants affected / at risk) | 28/136 | 34/164 | 24/114 | 29/137 | 21/100 | 19/120 | 26/91 | 22/121 | 18/85 | 18/119 | 15/80 | 14/115 | 15/79 | 18/113 | 12/79 | 12/109 | 9/74 | 8/104 | 10/68 | 12/102
Other Adverse Events (participants affected / at risk) | 104/136 | 136/164 | 90/114 | 103/137 | 80/100 | 93/120 | 68/91 | 81/121 | 65/85 | 77/119 | 57/80 | 71/115 | 51/79 | 71/113 | 52/79 | 63/109 | 50/74 | 60/104 | 37/68 | 55/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Week 1 (N=136) | Varenicline - Week 1 (N=164) | Placebo - Week 3 (N=114) | Varenicline - Week 3 (N=137) | Placebo - Week 4 (N=100) | Varenicline - Week 4 (N=120) | Placebo - Week 6 (N=91) | Varenicline - Week 6 (N=121) | Placebo - Week 7 (N=85) | Varenicline - Week 7 (N=119) | Placebo - Week 8 (N=80) | Varenicline - Week 8 (N=115) | Placebo - Week 10 (N=79) | Varenicline - Week 10 (N=113) | Placebo - Week 12 (N=79) | Varenicline - Week 12 (N=109) | Placebo - Week 14 (N=74) | Varenicline - Week 14 (N=104) | Placebo - Week 27 (N=68) | Varenicline - Week 27 (N=102)
Depressed Mood (Psychiatric disorders) | 3 | 3 | 3 | 4 | 2 | 4 | 1 | 6 | 1 | 4 | 4 | 4 | 0 | 2 | 0 | 4 | 1 | 2 | 0 | 0
Suicidal thoughts or i deation (Psychiatric disorders) | 4 | 15 | 6 | 8 | 3 | 6 | 9 | 6 | 5 | 7 | 5 | 4 | 3 | 5 | 3 | 2 | 3 | 1 | 1 | 5
Anxiety (Psychiatric disorders) | 5 | 3 | 1 | 3 | 1 | 4 | 2 | 5 | 1 | 3 | 2 | 1 | 3 | 3 | 3 | 2 | 0 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 20 | 19 | 10 | 16 | 12 | 10 | 12 | 9 | 10 | 11 | 7 | 10 | 8 | 10 | 9 | 7 | 5 | 7 | 8 | 4
Hostility (Psychiatric disorders) | 6 | 8 | 5 | 2 | 8 | 4 | 4 | 5 | 6 | 4 | 7 | 3 | 5 | 5 | 4 | 5 | 4 | 3 | 1 | 3
Irritability (Psychiatric disorders) | 4 | 1 | 3 | 3 | 4 | 3 | 5 | 4 | 3 | 3 | 2 | 1 | 2 | 5 | 1 | 1 | 2 | 2 | 2 | 1
Nausea (General disorders) | 0 | 1 | 2 | 3 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Headache (General disorders) | 1 | 3 | 2 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 1
Dizziness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in Attention (Psychiatric disorders) | 2 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Skin swelling or rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
skin redness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weakness on one or both sides of the body (General disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irregular heartbeat (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased heart rate (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Week 1 (N=136) | Varenicline - Week 1 (N=164) | Placebo - Week 3 (N=114) | Varenicline - Week 3 (N=137) | Placebo - Week 4 (N=100) | Varenicline - Week 4 (N=120) | Placebo - Week 6 (N=91) | Varenicline - Week 6 (N=121) | Placebo - Week 7 (N=85) | Varenicline - Week 7 (N=119) | Placebo - Week 8 (N=80) | Varenicline - Week 8 (N=115) | Placebo - Week 10 (N=79) | Varenicline - Week 10 (N=113) | Placebo - Week 12 (N=79) | Varenicline - Week 12 (N=109) | Placebo - Week 14 (N=74) | Varenicline - Week 14 (N=104) | Placebo - Week 27 (N=68) | Varenicline - Week 27 (N=102)
Nausea (General disorders) | 3 | 7 | 6 | 7 | 6 | 9 | 6 | 6 | 7 | 7 | 5 | 4 | 10 | 1 | 3 | 3 | 1 | 3 | 2 | 5
Abdominal Pain (Gastrointestinal disorders) | 21 | 23 | 13 | 28 | 14 | 28 | 15 | 24 | 14 | 21 | 12 | 21 | 12 | 21 | 15 | 15 | 13 | 11 | 8 | 17
Increased Flatulence (Gastrointestinal disorders) | 10 | 6 | 5 | 8 | 7 | 10 | 10 | 16 | 5 | 11 | 5 | 11 | 3 | 11 | 6 | 5 | 6 | 9 | 4 | 4
Constipation (Gastrointestinal disorders) | 6 | 5 | 3 | 4 | 5 | 5 | 7 | 10 | 3 | 8 | 5 | 8 | 3 | 9 | 4 | 4 | 5 | 5 | 3 | 6
Sleep problems (Psychiatric disorders) | 36 | 61 | 23 | 32 | 16 | 23 | 20 | 13 | 14 | 21 | 17 | 22 | 8 | 14 | 8 | 13 | 7 | 13 | 8 | 10
Insomnia (Psychiatric disorders) | 21 | 37 | 12 | 20 | 12 | 10 | 10 | 14 | 12 | 11 | 8 | 12 | 7 | 8 | 10 | 5 | 7 | 7 | 8 | 8
Abnormal Dreams (Psychiatric disorders) | 8 | 4 | 5 | 8 | 6 | 10 | 7 | 7 | 6 | 13 | 5 | 5 | 3 | 7 | 9 | 5 | 5 | 4 | 3 | 3
Irritability (Psychiatric disorders) | 16 | 30 | 11 | 14 | 12 | 15 | 8 | 16 | 11 | 10 | 12 | 14 | 11 | 10 | 6 | 8 | 7 | 6 | 3 | 7
Irregular Heartbeat (Cardiac disorders) | 1 | 6 | 0 | 2 | 3 | 3 | 4 | 3 | 2 | 6 | 1 | 3 | 1 | 4 | 1 | 3 | 2 | 3 | 0 | 0
Depressed Mood (Psychiatric disorders) | 37 | 41 | 15 | 21 | 19 | 16 | 9 | 14 | 13 | 17 | 8 | 16 | 15 | 15 | 10 | 6 | 7 | 7 | 9 | 15
Increased heart rate or palpitations (Cardiac disorders) | 7 | 19 | 7 | 8 | 5 | 13 | 7 | 13 | 4 | 13 | 4 | 11 | 4 | 10 | 5 | 10 | 3 | 8 | 2 | 3
Vomiting (General disorders) | 8 | 10 | 3 | 9 | 3 | 7 | 3 | 2 | 3 | 4 | 2 | 4 | 1 | 6 | 5 | 3 | 2 | 2 | 2 | 2
Dry Mouth (General disorders) | 10 | 16 | 9 | 13 | 11 | 17 | 5 | 10 | 6 | 12 | 4 | 7 | 3 | 7 | 5 | 5 | 7 | 1 | 3 | 2
Gastroesophageal reflux or indigestion (Gastrointestinal disorders) | 6 | 10 | 4 | 11 | 9 | 7 | 7 | 9 | 8 | 11 | 3 | 7 | 4 | 7 | 3 | 5 | 5 | 6 | 3 | 7
Anxiety (Psychiatric disorders) | 67 | 76 | 57 | 55 | 50 | 43 | 42 | 42 | 39 | 42 | 41 | 39 | 33 | 31 | 30 | 33 | 32 | 27 | 25 | 30
Skin swelling or rash (General disorders) | 10 | 7 | 7 | 1 | 7 | 6 | 5 | 6 | 4 | 5 | 6 | 3 | 4 | 3 | 5 | 0 | 8 | 5 | 3 | 4
Agitation (Psychiatric disorders) | 33 | 44 | 29 | 30 | 31 | 34 | 23 | 29 | 20 | 28 | 21 | 20 | 24 | 17 | 20 | 19 | 21 | 17 | 14 | 20
Headache (General disorders) | 6 | 15 | 8 | 9 | 7 | 7 | 8 | 9 | 4 | 10 | 4 | 5 | 1 | 5 | 4 | 5 | 1 | 5 | 3 | 5
Disturbance in attention (Psychiatric disorders) | 13 | 20 | 10 | 8 | 8 | 7 | 6 | 7 | 8 | 8 | 5 | 12 | 6 | 10 | 1 | 5 | 7 | 6 | 6 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dizziness (General disorders) | 15 | 20 | 9 | 17 | 11 | 9 | 11 | 12 | 10 | 13 | 7 | 11 | 6 | 11 | 6 | 6 | 8 | 4 | 4 | 9
Fatigue/lethargy (General disorders) | 36 | 41 | 20 | 20 | 18 | 23 | 15 | 18 | 15 | 13 | 7 | 17 | 12 | 13 | 7 | 12 | 9 | 11 | 6 | 10
Feeling of weakness without loss of strength (General disorders) | 12 | 14 | 4 | 6 | 7 | 7 | 4 | 8 | 3 | 4 | 2 | 3 | 1 | 4 | 0 | 6 | 4 | 3 | 2 | 2
Skin redness (General disorders) | 9 | 6 | 5 | 4 | 4 | 5 | 5 | 2 | 3 | 2 | 4 | 2 | 3 | 2 | 6 | 2 | 7 | 5 | 4 | 2
Hostility (Psychiatric disorders) | 17 | 21 | 14 | 11 | 12 | 14 | 5 | 12 | 9 | 18 | 8 | 13 | 14 | 11 | 10 | 11 | 9 | 9 | 10 | 8
Chest pain (General disorders) | 2 | 7 | 7 | 4 | 9 | 2 | 4 | 3 | 4 | 7 | 3 | 3 | 3 | 1 | 4 | 2 | 3 | 2 | 1 | 4
Weakness on one or both sides of the body (General disorders) | 21 | 23 | 18 | 14 | 9 | 10 | 7 | 9 | 9 | 15 | 6 | 10 | 7 | 11 | 6 | 13 | 10 | 10 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT02378714/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT02378714/ICF_001.pdf